CLINICAL TRIAL: NCT02997228
Title: Colorectal Cancer Metastatic dMMR/MSI-H Immuno-Therapy (COMMIT) Study: A Randomized Phase III Study of mFOLFOX6/Bevacizumab/Atezolizumab Combination Versus Single Agent Atezolizumab in the First-Line Treatment of Patients With Deficient DNA Mismatch Repair (dMMR)/Microsatellite Instability-High (MSI-H) Metastatic Colorectal Cancer
Brief Title: Testing the Addition of Atezolizumab to Combination Chemotherapy or Atezolizumab Alone for Metastatic Colon or Rectal Cancer, the COMMIT Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01961; NCI-2016-01961 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GI004/S1610; NRG-GI004 (Other: NRG Oncology); NRG-GI004 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2016-12-19; First posted 2016-12-20 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Colorectal Adenocarcinoma; Stage IV Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms | interventions — atezolizumab; Bevacizumab; Immunoglobulin G; Disulfides; Specimen Handling; Fluorouracil; dehydroftorafur; Leucovorin; Magnetic Resonance Spectroscopy; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (bevacizumab, mFOLFOX6) (Active Comparator): Patients receive bevacizumab intravenously (IV) over 30-90 minutes on day 1, oxaliplatin IV over 2 hours on day 1 of cycles 1-10, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1 and 2. Treatment with oxaliplatin repeats every 2 weeks for up to 10 cycles in the absence of disease progression or unacceptable toxicity. Treatment of bevacizumab, leucovorin calcium, and fluorouracil repeat every 2 weeks for up to 48 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT with or without PET or MRI throughout the trial. Patients may also undergo collection of optional blood samples throughout the trial. (CLOSED TO ACCRUAL)
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Leucovorin; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (atezolizumab) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1. Treatment repeats every 2 weeks for up to 48 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT with or without PET or MRI throughout the trial. Patients may also undergo collection of optional blood samples throughout the trial.
  Interventions: Drug: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (atezolizumab, bevacizumab, mFOLFOX6) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1. Treatment repeats every 2 weeks for up to 48 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive bevacizumab IV over 30-90 minutes on day 1, oxaliplatin IV over 2 hours on day 1 cycles 1-10, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV over 46-48 hours on day 1. Treatment with oxaliplatin repeats every 2 weeks for up to 10 cycles in the absence of disease progression or unacceptable toxicity. Treatment of bevacizumab, leucovorin calcium, and fluorouracil repeat every 2 weeks for up to 48 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT with or without PET or MRI throughout the trial. Patients may also undergo collection of optional blood samples throughout the trial.
  Interventions: Drug: Atezolizumab; Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Leucovorin; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm II (atezolizumab); Arm III (atezolizumab, bevacizumab, mFOLFOX6)
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm I (bevacizumab, mFOLFOX6); Arm III (atezolizumab, bevacizumab, mFOLFOX6)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or CT/PET
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm I (bevacizumab, mFOLFOX6); Arm III (atezolizumab, bevacizumab, mFOLFOX6)
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
  Arms: Arm I (bevacizumab, mFOLFOX6); Arm III (atezolizumab, bevacizumab, mFOLFOX6)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
  Arms: Arm I (bevacizumab, mFOLFOX6); Arm III (atezolizumab, bevacizumab, mFOLFOX6)
Procedure: Positron Emission Tomography — Undergo CT/PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well combination chemotherapy, bevacizumab, and/or atezolizumab work in treating patients with deficient deoxyribonucleic acid (DNA) mismatch repair colorectal cancer that has spread from where it first started (primary site) to other places in the body (metastatic). Chemotherapy drugs, such as fluorouracil, oxaliplatin, and leucovorin calcium, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of the tumor. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving combination chemotherapy, bevacizumab, and atezolizumab may work better in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy, based on progression-free survival (PFS), of fluorouracil, oxaliplatin, and leucovorin calcium (modified [m]FOLFOX6)/bevacizumab plus atezolizumab (combination) as compared to single agent atezolizumab.

SECONDARY OBJECTIVES:

I. To compare the overall survival. II. To compare the objective response rates (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

III. To determine the safety profiles of single agent atezolizumab and the combination of mFOLFOX6/bevacizumab/atezolizumab in patients with mismatch-repair deficient (dMMR)/microsatellite instability-high (MSI-H) metastatic colorectal cancer (mCRC).

IV. To determine the duration of response. V. To determine the duration of stable disease. VI. To determine the rate of progression-free survival (PFS) at 12 months. VII. To evaluate the disease control rate (complete response [CR] + partial response [PR] + stable disease [SD]) at 12 months.

TRANSLATIONAL OBJECTIVE:

I. To bank tissue and blood samples for other future correlative studies from patients enrolled on the study.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I (CLOSED TO ACCRUAL 6/4/2020): Patients receive bevacizumab intravenously (IV) over 30-90 minutes on day 1, oxaliplatin IV over 2 hours on day 1 of cycles 1-10, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1 and 2. Treatment with oxaliplatin repeats every 2 weeks for up to 10 cycles in the absence of disease progression or unacceptable toxicity. Treatment of bevacizumab, leucovorin calcium, and fluorouracil repeat every 2 weeks for up to 48 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) with or without positron emission tomography (PET) or magnetic resonance imaging (MRI) throughout the trial. Patients may also undergo collection of optional blood samples throughout the trial.

ARM II: Patients receive atezolizumab IV over 30-60 minutes on day 1. Treatment repeats every 2 weeks for up to 48 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT with or without PET or MRI throughout the trial. Patients may also undergo collection of optional blood samples throughout the trial.

ARM III: Patients receive atezolizumab IV over 30-60 minutes on day 1. Treatment repeats every 2 weeks for up to 48 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive bevacizumab IV over 30-90 minutes on day 1, oxaliplatin IV over 2 hours on day 1 cycles 1-10, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV over 46-48 hours on day 1. Treatment with oxaliplatin repeats every 2 weeks for up to 10 cycles in the absence of disease progression or unacceptable toxicity. Treatment of bevacizumab, leucovorin calcium, and fluorouracil repeat every 2 weeks for up to 48 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT with or without PET or MRI throughout the trial. Patients may also undergo collection of optional blood samples throughout the trial.

After completion of study treatment, patients are followed up every 8 weeks for 18 months, and then every 12 weeks for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have signed and dated an Institutional Review Board (IRB)-approved consent form that conforms to federal and institutional guidelines
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Diagnosis of metastatic adenocarcinoma of colon or rectum without previous chemotherapy or any other systemic therapy for metastatic colorectal cancer except for one cycle of FOLFOX or capecitabine and oxaliplatin (CAPOX), either with or without bevacizumab prior to enrollment. Upon enrollment, the preceding single cycle of FOLFOX or FOLFOX + bevacizumab, if the patient received one, will not count towards patients' assessments per protocol. Cycle 1 day 1 (C1D1) of atezolizumab or C1D1 of mFOLFOX6/bevacizumab + atezolizumab will correspond to the first day the patient received therapy on trial
* Tumor determined to be mismatch-repair deficient (dMMR) by Clinical Laboratory Improvement Act (CLIA)-certified immunohistochemical (IHC) assay with a panel of all four IHC markers, including MLH1, MSH2, PMS2, and MSH6; alternatively, MSI-H diagnosed by polymerase chain reaction (PCR)-based assessment of microsatellite alterations (either Bethesda markers or Pentaplex panel) or by next-generation sequencing (NGS) are eligible
* Documentation by PET/CT scan, CT scan, or MRI that the patient has measurable metastatic disease per RECIST 1.1
* No immediate need for surgical intervention for the primary tumor or palliative diversion/bypass
* Absolute neutrophil count (ANC) must be >= 1500/mm^3 (obtained within 28 days prior randomization)
* Platelet count must be >= 100,000/mm^3 (obtained within 28 days prior randomization)
* Hemoglobin must be >= 8 g/dL (obtained within 28 days prior randomization)
* Total bilirubin must be =< 4 x ULN (upper limit of normal) (obtained within 28 days prior randomization); and
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be =< 3 x ULN for the lab with the following exception: for patients with documented liver metastases, AST and ALT must be =< 5 x ULN (obtained within 28 days prior randomization)
* Calculated creatinine clearance >= 30 mL/min (obtained within 28 days prior randomization)
* A urine sample tested for proteinuria by either the dipstick method, urinalysis (UA), or a urine protein creatinine (UPC) ratio:

  * The dipstick method must indicate 0-1+ protein; if dipstick reading is >= 2+, a 24-hour urine must be done and it must demonstrate < 1.0 g of protein per 24 hours or a UPC ratio < 1.0
  * A urine protein creatinine (UPC) ratio must be < 1.0; if the UPC ratio is >= 1.0 a 24-hour urine must be done and it must demonstrate < 1.0 g of protein per 24 hours
  * Urinalysis must indicate < 30 mg/dl. If urinalysis >= 30 mg/dl, a 24-hour urine must be done and it must demonstrate < 1.0 g of protein per 24 hours or a UPC ratio < 1.0
* International normalized ratio of prothrombin time (INR) and prothrombin time (PT) must be =< 1.5 x ULN for the lab within 28 days before randomization; patients who are therapeutically treated with an agent such as warfarin may participate if they are on a stable dose and no underlying abnormality in coagulation parameters exists per medical history, regardless of PT/INR results
* Pregnancy test done within 28 days prior randomization must be negative (for women of childbearing potential only); pregnancy testing should be performed according to institutional standards; administration of atezolizumab or mFOLFOX6/bevacizumab/atezolizumab may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Women of child-bearing potential and men must agree to use adequate contraception methods that result in a failure rate of < 1% per year during the treatment period (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of atezolizumab, 6 months after the last dose of bevacizumab, and 6 months after the last dose of mFOLFOX6; a woman is considered to be of childbearing potential if she is not postmenopausal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus); examples of contraceptive methods with a failure rate of < 1% per year include: bilateral tubal ligation; male partner sterilization; intrauterine devices; the reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception; men must refrain from donating sperm during this same period

Exclusion Criteria:

* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies, fluoropyrimidines, folic acid derivatives or oxaliplatin
* Uncontrolled high blood pressure defined as systolic blood pressure (BP) > 150 mmHg or diastolic BP > 100 mmHg with or without anti-hypertensive medication; patients with initial BP elevations are eligible if initiation or adjustment of BP medication lowers pressure to meet entry criteria
* Documented New York Heart Association (NYHA) class III or IV congestive heart failure
* Serious or non-healing wound, skin ulcer, or bone fracture
* History of inherited bleeding diathesis, gastrointestinal (GI) perforation, significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis or symptomatic peripheral ischemia, transient ischemic attack [TIA], cerebrovascular accident [CVA] or arterial thrombotic event), abdominal fistula, intra-abdominal abscess, or active GI bleeding (with cause not addressed) within 6 months prior to randomization, or other medical condition in the opinion of the treating oncologist that makes the risk of cardiovascular or bleeding complications with bevacizumab use unacceptably high
* Other malignancies are excluded unless the patient has completed therapy for the malignancy >= 12 months prior to randomization and is considered disease-free; patients with the following cancers are eligible if diagnosed and treated within the past 12 months: in situ carcinomas or basal cell and squamous cell carcinoma of the skin
* Known DPD (dihydro pyrimidine dehydrogenase) deficiency
* Symptomatic peripheral sensory neuropathy >= grade 2 (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0)
* Prior treatment with oxaliplatin chemotherapy within 6 months prior to randomization
* History of grade 2 hemoptysis (defined as 2.5 mL of bright red blood per episode) within 1 month prior to screening
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents; patients who have received prior treatment with anti-CTLA-4 may be enrolled provided the following requirements are met:

  * Minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose to randomization
  * No history of severe immune-related adverse effects (CTCAE grade 3 and 4) from anti-CTLA-4
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 14 days prior to randomization; however,

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea; or chronic daily treatment with corticosteroids with a dose of =< 10 mg/day methylprednisolone equivalent) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease; however,

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HbsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible if polymerase chain reaction (PCR) for hepatits B virus (HBV) ribonucleic acid (RNA) is negative per local guidelines
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA per local guidelines
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis; however,

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or active or recently active (within 90 days of randomization) pneumonitis (including drug induced) that required systemic immunosuppressive therapy (i.e. corticosteroids, etc.). History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients with known active tuberculosis (TB) are excluded
* Severe infections within 28 days prior to randomization, including but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 14 days prior to randomization
* Received oral or intravenous (IV) antibiotics within 14 days prior to randomization; patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization or anticipation of need for a major surgical procedure during the course of the study
* The administration of a live, attenuated vaccine within 28 days prior to randomization
* Pregnant women are excluded from this study because atezolizumab is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with atezolizumab, breastfeeding should be discontinued if the mother is treated with atezolizumab; these potential risks may also apply to other agents used in this study; (Note: pregnancy testing should be performed within 28 days prior to randomization according to institutional standards for women of childbearing potential)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-19 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From the time from randomization until first confirmed progression or death from any cause, assessed up to 5 years
  The analysis set is intent-to-treat (ITT). The experimental arms will be compared to the control arm by the log-rank test stratified by BRAF status (V600E mutation or not), metastatic disease: (liver-only, extra-hepatic), and prior adjuvant therapy for colon cancer (yes, no). Hazard ratios and associated confidence intervals from a stratified Cox regression model will also be reported along with estimates of the distributions of time to PFS event by the method of Kaplan and Meier. Sensitivity analyses accounting for 2 or more consecutively missed scheduled tumor imaging scans before progression/death will also be conducted.

SECONDARY OUTCOMES:
Overall survival (OS) | The time from randomization to death from any cause, assessed up to 5 years
  Will be analyzed using the stratified log rank test and the ITT population. Kaplan-Meier plots will illustrate the distribution of these endpoints by treatment. Stratified Cox regression models will be used to estimate hazard ratios and associated confidence intervals.
Objective response rate (ORR) (complete response [CR] or partial response [PR]) | Up to 5 years
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Will be analyzed by a logistic regression models that control for the stratification factors (BRAF status, liver involvement, and adjuvant chemotherapy [chemo]) using the ITT population. Observed proportions along with confidence intervals will be presented by treatment.
Incidence of adverse events | Up to 30 days after last cycle
  Defined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The safety profile will be described by tabulating the maximum observed grade of adverse event for each individual adverse event, for each system organ class, and overall using the Safety population.
Rate of PFS | At 12 months
Disease control rate (CR + PR + stable disease [SD]) | At 12 months
  Assessed by RECIST 1.1. Will be analyzed by a logistic regression models that control for the stratification factors (BRAF status, liver involvement, and adjuvant chemo) using the ITT population. Observed proportions along with confidence intervals will be presented by treatment.
Duration of overall response (CR or PR) | From the time of first response to first confirmed progression by the study investigator or death from any cause, assessed up to 5 years
  Assessed by RECIST 1.1. Will be analyzed using the stratified log rank test and the ITT population. Kaplan-Meier plots will illustrate the distribution of these endpoints by treatment. Stratified Cox regression models will be used to estimate hazard ratios and associated confidence intervals.
Duration of SD | From the time of first on-study assessment of SD to first progression by the study investigator or death from any cause, assessed up to 5 years
  Assessed per RECIST 1.1. Will be analyzed using the stratified log rank test and the ITT population. Kaplan-Meier plots will illustrate the distribution of these endpoints by treatment. Stratified Cox regression models will be used to estimate hazard ratios and associated confidence intervals.

OTHER OUTCOMES:
Severity of fatigue | At 16 weeks
  Will use the ITT population. Measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue questionnaire. Will be compared between the control arm (Chemo-bevacizumab [Bev]) and the experimental arm by means of ordinal logistic regression with adjustment for the corresponding baseline measurement and stratification variables. The comparison will be performed at the significance level of 0.05 (two-sided) and the clinical meaningfulness of the comparison will be considered.
Physical functioning | At 16 weeks
  Will use the ITT population. Measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality-of-Life questionnaire (QLQ)-C30 physical functioning scale. Will be compared between the control arm (Chemo-Bev) and the experimental arm by means of ordinal logistic regression with adjustment for the corresponding baseline measurement and stratification variables. The comparison will be performed at the significance level of 0.05 (two-sided) and the clinical meaningfulness of the comparison will be considered.
Health utility scores | Up to 5 years
  Will use the ITT population. Will be measured using the EuroQoL 5 Dimensions 5 Levels (EQ-5D-5L) questionnaire.
Proportion of patients reporting each response option at each assessment timepoint by treatment arm for item GP5 from the Functional Assessment of Cancer Therapy - General (FACT-G) | Up to 5 years
  Will use the ITT population.
Intratumoral lymphocyte PD-L1+ expression (>= 1 % is positive) by immunohistochemistry (IHC) as a predictive biomarker of efficacy | Up to 5 years
  Will use the ITT population.
Efficacy dependent on the number of somatic mutations | Up to 5 years
  Will use the ITT population.
Efficacy in tumors with MLH1 silencing | Up to 5 years
  Will use the ITT population.
Change in quantification of cell free deoxyribonucleic acid (cfDNA) mutations | Baseline up to 5 years
  Will use the ITT population.
Development of progression or relapse to treatment in cfDNA | Up to 5 years
  Will use the ITT population.
Changes in T-cell repertoire diversity as a predictive biomarker of efficacy | Baseline up to 5 years
  Will use the ITT population.
PFS of patients with high levels of diversity | Up to 5 years
  Compared to patients with low levels of diversity. Will use the ITT population.
Change in T-cell diversity | Baseline to first restaging between immunotherapy arms and the standard of care arm
  Will use the ITT population.
Mechanism of immune resistance to PD-1 blockade in mismatch repair deficient (dMMR)/microsatellite instability-high metastatic colorectal cancer (mCRC) by comparative analysis of tumor samples collected | Baseline up to 5 years
  Will use the ITT population.

CONTACTS AND LOCATIONS:
Overall Officials: Caio Max S Rocha Lima, Principal Investigator — NRG Oncology
Locations (446):
- United States (446):
  - Kingman Regional Medical Center, Kingman, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - John Muir Medical Center-Concord, Concord, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - William Backus Hospital, Norwich, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta Oncology Associates PC-Wheeler, Augusta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Franciscan Saint Elizabeth Health - Lafayette East, Lafayette, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - HaysMed, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Norton Audubon Hospital and Medical Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente Lutherville - Timonium Medical Center, Lutherville, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - McLaren Cancer Institute-Bloomfield, Bloomfield, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Rochester, Rochester, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Saint Luke's Hospital-Quakertown Campus, Quakertown, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Baptist Hospitals of Southeast Texas Cancer Center, Beaumont, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - STCC at DHR Health Institute for Research and Development, Edinburg, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Baptist Regional Cancer Network-Cancer Center of Southeast Texas, Port Arthur, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Kaiser Permanente-Caton Hill Medical Center, Woodbridge, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming